CLINICAL TRIAL: NCT06677658
Title: Effects of Olive Oil on Clinical, Laboratory and Survival in Patients Given Pulse Steroid Treatment for Covid-19 Pneumonia
Brief Title: The Role of Olive Oil in the Treatment of Covid-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Other Study IDs: 22.05.2024-03
Record Dates: First submitted 2024-11-02; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: COVID-19 Pneumonia; Nutrition, Healthy
Keywords: COVID-19; Pneumonia; Olive Oil; Steroid; Immune system
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Olive Oil; Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients diagnosed with COVID-19 pneumonia treated with pulse steroids (250 mg/day) for three days and routinely consumed at least 20 ml/day olive oil in their diets were defined as Group 1.
  Interventions: Dietary Supplement: Olive Oil; Drug: Methylprednisolone
- Group 2: Patients of similar age and gender with COVID-19 pneumonia who received the same treatment but did not consume olive oil were defined as Group 2.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Dietary Supplement: Olive Oil — Group 1 included patients who consumed at least 20 ml of oral olive oil daily. Group 2 included patients who did not consume olive oil.
  Groups: Group 1
Drug: Methylprednisolone — Both groups were diagnosed with Covid-19 pneumonia and were given pulse steroid ( methylprednisolone ) treatment at 250 mg/day for 3 days.
  Other Names: Pulse steroid

SUMMARY:
Objective: Consuming natural olive oil in patients diagnosed with COVID-19 Pneumonia may strengthen immunity, slow down disease progression, and lower mortality. Within the scope of this research, the investigators aimed to elucidate the effect of using natural olive oil on clinical, laboratory, and radiological findings and survival in patients diagnosed with COVID-19 pneumonia and given pulse steroid treatment.

Method: This retrospective observational research enrolled 130 patients diagnosed with COVID-19 pneumonia. Participants were examined in two groups according to their olive oil consumption status. Patients diagnosed with COVID-19 pneumonia treated with pulse steroids for three days who routinely consumed oral olive oil in their daily diets were defined as Group 1, and those who did not consume olive oil were defined as Group 2.

DETAILED DESCRIPTION:
Introduction: In the COVID-19 pandemic, many patients with lung involvement who received pulse steroid treatment showed improvement in clinical, laboratory, radiological, and survival parameters. It was observed that a significant number of patients who showed improvement consumed natural olive oil, and while the follow-up and treatment of these patients continued, the effect of oral consumption of natural olive oil on clinical, laboratory parameters, and survival of the patients was the subject of research [1]. The benefits of olive oil consumption can be increased through physical activity, especially strength and resistance exercise. Such an approach is likely to prevent viral infections effectively. In terms of the recommended dose of olive oil, a moderate dose of 20-30 grams/day (especially extra virgin olive oil rich in polyphenols) can be recommended in combination with other dietary functional foods to strengthen the immune system, which is in line with the latest non-communicable disease prevention recommendations [1, 2]. The Mediterranean diet, which includes extra virgin olive oil and a correct lifestyle, can prevent low-grade inflammation and other chronic pathologies by directly affecting the intestinal microbiota and the immune system. A study has stated that olive oil can be used pharmacotherapeutically against SARS-CoV 2 [3]. In this context, it has been predicted that the consumption of natural olive oil in patients diagnosed with COVID-19 Pneumonia may strengthen immunity, slow down disease progression, and lower mortality. Within the scope of this research, we aimed to elucidate the effect of using natural olive oil on clinical, laboratory, and radiological findings and survival in patients diagnosed with COVID-19 pneumonia and given pulse steroid treatment.

Method: This retrospective observational research enrolled 130 patients diagnosed with COVID-19 pneumonia, confirmed with real-time polymerase chain reaction (RT-PCR). The patients were segmented into two groups (n=65 in each) according to their olive oil consumption. All procedures followed were in accordance with the ethical standards of the responsible committee on human experimentation (institutional and national) and with the Helsinki Declaration of 1975, as revised in 2008. Ethics committee approval has been granted from our institution with protocol number 22.05.2024/03, and informed consent has been obtained from all participants.

Participants were examined in two groups according to their olive oil consumption status. Patients diagnosed with COVID-19 pneumonia treated with pulse steroids ( methylprednisolone 250 mg/day) for three days and routinely consumed at least 20 ml olive oil in their daily diets were defined as Group 1. Patients of similar age and gender with COVID-19 pneumonia who received the same treatment but did not consume olive oil were defined as Group 2.

References:

1. Soo CI, Poon KV, Ayub A, You HW, Tan CX, Loh KJJ, et al. High-dose pulse methylprednisolone vs. dexamethasone standard therapy for severe and critical COVID-19 pneumonia: Efficacy assessment in a retrospective single-centre experience from Malaysia. Medical Journal of Malaysia. 2024;79(1):15-20.
2. Alkhatib A. Antiviral functional foods and exercise lifestyle prevention of coronavirus. Nutrients. 2020;12(9):2633. doi: 10.3390/nu12092633.
3. Hendi AA, Virk P, Awad MA, Elobeid M, Ortashi KM, Alanazi MM, et al. In silico studies on zinc oxide based nanostructured oil carriers with seed extracts of Nigella sativa and Pimpinella anisum as potential inhibitors of 3CL protease of SARS-CoV-2. Molecules. 2022;27(13):4301. doi: 10.3390/molecules27134301.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients aged ≥18 who were diagnosed with COVID-19 and had lung involvement (COVID-19 pneumonia).

Exclusion Criteria:

* Patients under the age of 18, pregnant women, individuals intubated due to severe respiratory failure in COVID-19 pneumonia, and those who received alternative treatments other than pulse steroid treatment (Immunoplasma, Tocilizumab, Anakinra, Plasmapheresis, Stem Cell Therapy, etc.) were excluded

Ages: 27 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research enrolled 130 patients diagnosed with COVID-19 pneumonia, confirmed with real-time polymerase chain reaction (RT-PCR). The patients were segmented into two groups (n=65 in each) according to their olive oil consumption. However, all of the patients included in the study were patients diagnosed with covid-19 pneumonia and given pulse steroid treatment.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Positive effect of olive oil on clinical and laboratory parameters in patients given pulse steroid therapy due to Covid 19 pneumonia. | After 3 days of 250 mg/day pulse steroid ( methylprednisolone ) treatment and during hospital stay.
  The benefits of olive oil consumption can be increased through physical activity, especially strength and resistance exercise. Such an approach is likely to prevent viral infections effectively. In terms of the recommended dose of olive oil, a moderate dose of 20-30 grams/day (especially extra virgin olive oil rich in polyphenols) can be recommended in combination with other dietary functional foods to strengthen the immune system, which is in line with the latest non-communicable disease prevention recommendations.
  Positive effects of regular daily olive oil use on clinical and laboratory parameters were observed in patients receiving pulse steroid treatment due to Covid-19 pneumonia.

SECONDARY OUTCOMES:
Intensive care requirement and mortality in patients diagnosed with covid-19 pneumonia taking olive oil. | After 3 days of 250 mg/day pulse steroid treatment and during hospital stay
  Among patients diagnosed with Covid-19 pneumonia and given pulse steroid treatment, those who routinely used olive oil in their daily diets required less intensive care and had lower mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Günaydın, MD, Study Chair — Assistant researcher; Ersin Kuloğlu, MD, Study Chair — Assistant researcher; Gökhan Aydın, MD, Study Chair — Assistant researcher
Locations (1):
- Giresun Training and Research Hospital, Giresun, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soo CI, Poon KV, Ayub A, You HW, Tan CX, Loh KJJ, Eng CCH, Sia LC, Wong CK. High-dose pulse methylprednisolone vs. dexamethasone standard therapy for severe and critical COVID-19 pneumonia: Efficacy assessment in a retrospective single-centre experience from Malaysia. Med J Malaysia. 2024 Jan;79(1):15-20. PMID 38287752
- [Background] Alkhatib A. Antiviral Functional Foods and Exercise Lifestyle Prevention of Coronavirus. Nutrients. 2020 Aug 28;12(9):2633. doi: 10.3390/nu12092633. PMID 32872374
- [Background] Hendi AA, Virk P, Awad MA, Elobeid M, Ortashi KMO, Alanazi MM, Alkallas FH, Almoneef MM, Abdou MA. In Silico Studies on Zinc Oxide Based Nanostructured Oil Carriers with Seed Extracts of Nigella sativa and Pimpinella anisum as Potential Inhibitors of 3CL Protease of SARS-CoV-2. Molecules. 2022 Jul 4;27(13):4301. doi: 10.3390/molecules27134301. PMID 35807545